CLINICAL TRIAL: NCT07182799
Title: Definition of Intra-procedural Optical Coherence Tomography (OCT) Clinical Impact, Both in Terms of Revascularization Indication and Procedural Result.
Brief Title: Starring Optical Coherence Tomography During Percutaneous Coronary Intervention Guidance
Acronym: OCT-AGEM
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Romagnoli Enrico, Clinical Physician, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7262
Record Dates: First submitted 2025-09-02; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndromes (ACS); Chronic Coronary Syndrome; MINOCA; INOCA (Ischemia With Non Obstructive Coronary Artery Disease); Percutaneous Coronary Intervention (PCI); Coronary Stent Implantation; Stent Restenosis; Stent Thrombosis; Clinical Outcome
Keywords: Percutaneous coronary intervention; Optical Coherence Tomography; Acute coronary syndrome; Chronic coronary syndrome; Clinical outcome; Coronary plaque; Coronary stent optimization
MeSH Terms: conditions — Acute Coronary Syndrome; MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-interventional: Patients undergoing an OCT coronary assessment during a clinically indicated coronary angiogram, resulting in a non-obstructive coronary artery disease
  Interventions: Diagnostic Test: Plaque vulnerability assessment
- Interventional: Patients undergoing an OCT coronary assessment during a clinically indicated coronary angiogram, guiding a percutaneous coronary intervention
  Interventions: Diagnostic Test: Stent implantation optimization

INTERVENTIONS:
Diagnostic Test: Plaque vulnerability assessment — The purpose of the OCT-AGEM registry is to confirm the clinical utility of plaque OCT assessment over the standard coronary angiography evaluation. In particular, this ambispective cohort study aims to validate the predictive value of the OCT-based plaque vulnerability criteria:
  * Minimum lumen area <3.5 mm2;
  * Fibrous cap minimum thickness <65 µm;
  * Lipid arc extension >180°;
  * Presence of macrophages;
  * Superficial and deep calcified nodules
  * Ulceration/Erosion/Dissection
  * Layered tissue
  * Optical flow ratio (OFR)
  Other Names: Minimum lumen area; Fibrous cap minimum thickness; Lipid arc extension; Presence of macrophages; Superficial and deep calcified nodules; Ulceration/Erosion/Dissection; Layered tissue; Plaque burden (%); Optical flow ratio (OFR)
  Groups: Non-interventional
Diagnostic Test: Stent implantation optimization — The purpose of the OCT-AGEM registry is to confirm the clinical utility of OCT guidance during PCI over the standard coronary angiography evaluation. In particular, this ambispective cohort study aims to validate the predictive value of the OCT-derived plaque/stent parameters reported in expert consensus OCT documents, utilizing the cut-off points identified in the previous OCT registries
  Other Names: Minimum lumen area; Fibrous cap minimum thickness; Lipid arc extension; Presence of macrophages; Superficial and deep calcified nodules; Ulceration/Erosion/Dissection; Layered tissue; Plaque burden (%); Stent edge dissection; Reference narrowing; Stent malapposition; Minimum stent area; Stent expansion (%); In-stent tissue protrusion; Stent deformation; Stent geometry; Neo-carina shaping; Optical flow ratio (OFR)
  Groups: Interventional

SUMMARY:
The starring optical coherence tomography during percutaneous coronary intervention guidance (OCT-AGEM) registry aims to evaluate the clinical impact of intra-procedural optical coherence tomography (OCT) in coronary revascularization, both in guiding revascularization decisions and optimizing interventional procedural outcomes, as well as assessing mid- and long-term clinical results.

DETAILED DESCRIPTION:
The OCT-AGEM registry is an ambispective, single-center observational cohort study comprising a retrospective registry (Phase I) and a prospective registry (Phase II). All patients aged 18 years or older undergoing OCT assessment during a clinically indicated coronary angiography, regardless of clinical presentation (silent ischemia, stable angina, or acute coronary syndrome), are eligible. The retrospective phase targets approximately 2,200 patients, while the prospective phase will enroll 1,000 patients, based on a current annual rate of about 150 OCT-guided procedures. Sample size calculations, informed by prior studies and preliminary experience, are as follows: for the non-interventional arm, assuming a 5% cumulative incidence of the composite endpoint and a 20% prevalence of OCT-defined vulnerable plaque, a total of 1,100 patients is required (hazard ratio [HR] 0.80; 80% power); for the interventional arm, assuming a 25% incidence of OCT-defined suboptimal stent implantation and 12% for the composite endpoint, a total of 2,100 patients will be enrolled (HR 0.85; 80% power). The study will investigate the predictive clinical value of OCT-defined vulnerable plaque in patients with non-obstructive coronary artery disease (MINOCA/INOCA) and the prognostic impact of OCT-derived plaque and stent parameters in patients undergoing percutaneous coronary intervention (PCI). The primary composite endpoint includes cardiac death, target-vessel myocardial infarction, target lesion revascularization, and stent thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Patients with clinical indication to coronary angiography undergoing intra-procedural OCT regardless of the clinical syndrome;
* Patients with at least one end-procedural OCT assessment with a sufficient acquisition length to address the whole length of plaque or stented segments plus the proximal and distal reference segments;
* Patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Female with childbearing potential or lactating;
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl and/or glomerular filtration rate <30 ml/min);
* Advanced heart failure (NYHA III-IV);
* Previous heart transplantation;
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study;
* Heavily calcified lesion or tortuous vessel which cannot be successfully imaged by OCT;
* Lesion located at the coronary ostium or in angulated (>70°), sharp take-off vessel;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects over 18 years who are undergoing an OCT coronary assessment during clinically indicated coronary angiogram regardless of the clinical syndrome (silent ischemia, effort angina or acute coronary syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2036-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cardiac death or target-vessel myocardial infarction or target lesion revascularization (non-interventional group) | 1 year, 3 years, and 5 years
  Composite outcome including cardiac death (i.e. any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death), target-vessel myocardial infarction (i.e. any spontaneous myocardial infarction attributed to the vessel studied with OCT), and target lesion revascularization (i.e. any target-lesion revascularization by means of percutaneous coronary intervention and coronary artery bypass grafting).
Number of patients with cardiac death or target-vessel myocardial infarction or target lesion revascularization or stent restenosis/thrombosis (interventional group) | 1 year, 3 years, and 5 years
  Composite outcome including cardiac death (i.e. any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death), target-vessel myocardial infarction (i.e. any spontaneous myocardial infarction attributed to the vessel studied with OCT), target lesion revascularization (i.e. any target-lesion revascularization by means of percutaneous coronary intervention and coronary artery bypass grafting), and stent restenosis (i.e. angiographic in-stent stenosis/thrombosis >50%).

SECONDARY OUTCOMES:
Predictive value of single vulnerable plaque OCT-derived criteria (non-interventional and interventional group) in terms of incidence of the primary and secondary outcomes | 1 year, 3 years, and 5 years
  Clinical impact of the single pre-specified OCT features of plaque vulnerability:
  * Minimum lumen area <3.5 mm2 (measured along the entire length of the assessed coronary segment );
  * Fibrous cap minimum thickness <65 µm (defined as a signal-rich homogeneous band overlying a lipid core, and measured at the thinnest portion);
  * Lipid arc extension >180° (defined as a signal-poor region diffusely bordered by overlying signal-rich bands corresponding to a fibrous cap);
  * Presence of macrophages (characterized at visual estimation as signal-rich, distinct, or confluent punctate regions that exceed the intensity of background speckle noise);
  * Superficial and deep calcified nodules (protruding mass with irregular surface characterized by signal-poor heterogeneous regions with sharp borders)
  * Ulceration/Erosion/Dissection (linear rim of tissue with a width ≥200μm and a clear separation from the vessel wall or underlying plaque)
  * Layered tissue (plaque with one or more evident layers)
Predictive clinical value of single pre-specified plaque/stent OCT features in patients undergoing percutaneous coronary revascularization (interventional group) in terms of incidence of the primary and secondary outcomes | 1 year, 3 years, and 5 years
  Clinical impact of the single pre-specified OCT features of the stented plaques:
  * Edge dissection with a width ≥200μm (linear rim of tissue with a width ≥200μm and a clear separation from the vessel wall or underlying plaque);
  * Reference narrowing: lumen area <4.5mm2 in the presence of significant residual plaque adjacent to stent endings (including 5mm beyond stent borders);
  * Malapposition >200μm (stent-adjacent vessel lumen distance >200μm);
  * In-stent minimum lumen area (MLA) <4.5mm2 (measure of smaller in-stent lumen area);
  * In-stent MLA <80% (expressed as % of the average reference lumen areas);
  * Intrastent plaque/thrombus protrusion ≥500μm in thickness (tissue prolapsing between stent struts extending inside a circular arc connecting adjacent struts or intraluminal mass ≥500μm in thickness with no direct continuity with the surface of the vessel wall or highly backscattered luminal protrusion in continuity with the vessel wall and resulting in signal-free shadowing).
Number of patients with cardiac death | 1 year, 3 years, and 5 years
  Cardiac death will be defined as any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death.
Number of patients with non-fatal spontaneous target-vessel myocardial infarction (excluding peri-procedural myocardial infarction) | 1 year, 3 years, and 5 years
  Any spontaneous myocardial infarction will be attributed to the target vessel if not clearly attributable to the non-target vessels.
Number of patients with target lesion revascularization | 1 year, 3 years, and 5 years
  Any lesion revascularization will be considered in case of percutaneous coronary intervention or coronary artery bypass grafting of the studied lesion.
Number of patients with restenosis or thrombosis of the target lesion | 1 year, 3 years, and 5 years
  Any revascularization procedure performed because of angiographic restenosis/thrombosis >50% at the site of the target lesion associated with clinical or objective evidence of inducible myocardial ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Romagnoli, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Francesco Burzotta, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prati F, Romagnoli E, Gatto L, La Manna A, Burzotta F, Limbruno U, Versaci F, Fabbiocchi F, Di Giorgio A, Marco V, Ramazzotti V, Di Vito L, Trani C, Porto I, Boi A, Tavazzi L, Mintz GS. Clinical Impact of Suboptimal Stenting and Residual Intrastent Plaque/Thrombus Protrusion in Patients With Acute Coronary Syndrome: The CLI-OPCI ACS Substudy (Centro per la Lotta Contro L'Infarto-Optimization of Percutaneous Coronary Intervention in Acute Coronary Syndrome). Circ Cardiovasc Interv. 2016 Dec;9(12):e003726. doi: 10.1161/CIRCINTERVENTIONS.115.003726. PMID 27965297
- [Background] Romagnoli E, Gatto L, La Manna A, Burzotta F, Taglieri N, Saia F, Amico F, Marco V, Ramazzotti V, Di Giorgio A, Di Vito L, Boi A, Contarini M, Castriota F, Mintz GS, Prati F. Role of residual acute stent malapposition in percutaneous coronary interventions. Catheter Cardiovasc Interv. 2017 Oct 1;90(4):566-575. doi: 10.1002/ccd.26974. Epub 2017 Mar 15. PMID 28295990
- [Background] Prati F, Romagnoli E, La Manna A, Burzotta F, Gatto L, Marco V, Fineschi M, Fabbiocchi F, Versaci F, Trani C, Tamburino C, Alfonso F, Mintz GS. Long-term consequences of optical coherence tomography findings during percutaneous coronary intervention: the Centro Per La Lotta Contro L'infarto - Optimization Of Percutaneous Coronary Intervention (CLI-OPCI) LATE study. EuroIntervention. 2018 Jul 20;14(4):e443-e451. doi: 10.4244/EIJ-D-17-01111. PMID 29633940
- [Background] Gatto L, Alfonso F, Paoletti G, Burzotta F, La Manna A, Budassi S, Biccire FG, Fineschi M, Marco V, Fabbiocchi F, Vergallo R, Boi A, Ruscica G, Versaci F, Taglieri N, Calligaris G, Albertucci M, Romagnoli E, Ramazzotti V, Tamburino C, Crea F, Ozaki Y, Arbustini E, Prati F. Relationship betweeen the amount and location of macrophages and clinical outcome: subanalysis of the CLIMA-study. Int J Cardiol. 2022 Jan 1;346:8-12. doi: 10.1016/j.ijcard.2021.11.042. Epub 2021 Nov 17. PMID 34798205
- [Background] Prati F, Romagnoli E, Biccire FG, Burzotta F, La Manna A, Budassi S, Ramazzotti V, Albertucci M, Fabbiocchi F, Sticchi A, Trani C, Calligaris G, Fineschi M, Versaci F, Tamburino C, Ozaki Y, Alfonso F, Mintz GS. Clinical outcomes of suboptimal stent deployment as assessed by optical coherence tomography: long-term results of the CLI-OPCI registry. EuroIntervention. 2022 Jun 3;18(2):e150-e157. doi: 10.4244/EIJ-D-21-00627. PMID 34825652
- [Background] Romagnoli E, Ramazzotti V, Burzotta F, Gatto L, Marco V, Paoletti G, Biondi-Zoccai G, Alfonso F, Crea F, Trani C, Prati F; CLI-OPCI Project Investigators*. Definition of Optimal Optical Coherence Tomography-Based Stent Expansion Criteria: In-Stent Minimum Lumen Area Versus Residual Stent Underexpansion. Circ Cardiovasc Interv. 2022 Sep;15(9):e011496. doi: 10.1161/CIRCINTERVENTIONS.121.011496. Epub 2022 Sep 20. PMID 36126136
- [Background] Romagnoli E, Burzotta F, Vergallo R, Gatto L, Biondi-Zoccai G, Ramazzotti V, Biccire F, Budassi S, Trani C, Ali Z, Stone GW, Prati F. Clinical impact of OCT-derived suboptimal stent implantation parameters and definitions. Eur Heart J Cardiovasc Imaging. 2023 Dec 21;25(1):48-57. doi: 10.1093/ehjci/jead172. PMID 37463223
- [Background] Biccire FG, Fabbiocchi F, Gatto L, La Manna A, Ozaki Y, Romagnoli E, Marco V, Boi A, Fineschi M, Piedimonte G, Cerrato E, Musto C, Taglieri N, Di Giorgio A, Vizzari G, Ruscica G, Canova PA, Vergallo R, Burzotta F, Limbruno U, Albertucci M, Raber L, Crea F, Alfonso F, Arbustini E, Stone GW, Prati F. Long-Term Prognostic Impact of OCT-Derived High-Risk Plaque Features: Extended Follow-Up of the CLIMA Study. JACC Cardiovasc Interv. 2025 Jun 9;18(11):1361-1372. doi: 10.1016/j.jcin.2025.04.044. PMID 40500004
- [Background] Tanigawa J, Barlis P, Di Mario C. Intravascular optical coherence tomography: optimisation of image acquisition and quantitative assessment of stent strut apposition. EuroIntervention. 2007 May;3(1):128-36. PMID 19737696
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Niccoli G, Montone RA, Di Vito L, Gramegna M, Refaat H, Scalone G, Leone AM, Trani C, Burzotta F, Porto I, Aurigemma C, Prati F, Crea F. Plaque rupture and intact fibrous cap assessed by optical coherence tomography portend different outcomes in patients with acute coronary syndrome. Eur Heart J. 2015 Jun 7;36(22):1377-84. doi: 10.1093/eurheartj/ehv029. Epub 2015 Feb 18. PMID 25713314
- [Background] Prati F, Uemura S, Souteyrand G, Virmani R, Motreff P, Di Vito L, Biondi-Zoccai G, Halperin J, Fuster V, Ozaki Y, Narula J. OCT-based diagnosis and management of STEMI associated with intact fibrous cap. JACC Cardiovasc Imaging. 2013 Mar;6(3):283-7. doi: 10.1016/j.jcmg.2012.12.007. PMID 23473109
- [Background] Souteyrand G, Arbustini E, Motreff P, Gatto L, Di Vito L, Marco V, Amabile N, Chisari A, Kodama T, Romagnoli E, Tavazzi L, Crea F, Narula J, Prati F. Serial optical coherence tomography imaging of ACS-causing culprit plaques. EuroIntervention. 2015 Jul;11(3):319-24. doi: 10.4244/EIJV11I3A59. PMID 26196754
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Prati F, Guagliumi G, Mintz GS, Costa M, Regar E, Akasaka T, Barlis P, Tearney GJ, Jang IK, Arbustini E, Bezerra HG, Ozaki Y, Bruining N, Dudek D, Radu M, Erglis A, Motreff P, Alfonso F, Toutouzas K, Gonzalo N, Tamburino C, Adriaenssens T, Pinto F, Serruys PW, Di Mario C; Expert's OCT Review Document. Expert review document part 2: methodology, terminology and clinical applications of optical coherence tomography for the assessment of interventional procedures. Eur Heart J. 2012 Oct;33(20):2513-20. doi: 10.1093/eurheartj/ehs095. Epub 2012 May 31. No abstract available. PMID 22653335
- [Background] Burzotta F, Leone AM, Aurigemma C, Zambrano A, Zimbardo G, Arioti M, Vergallo R, De Maria GL, Cerracchio E, Romagnoli E, Trani C, Crea F. Fractional Flow Reserve or Optical Coherence Tomography to Guide Management of Angiographically Intermediate Coronary Stenosis: A Single-Center Trial. JACC Cardiovasc Interv. 2020 Jan 13;13(1):49-58. doi: 10.1016/j.jcin.2019.09.034. PMID 31918942
- [Background] Prati F, Romagnoli E, Gatto L, La Manna A, Burzotta F, Ozaki Y, Marco V, Boi A, Fineschi M, Fabbiocchi F, Taglieri N, Niccoli G, Trani C, Versaci F, Calligaris G, Ruscica G, Di Giorgio A, Vergallo R, Albertucci M, Biondi-Zoccai G, Tamburino C, Crea F, Alfonso F, Arbustini E. Relationship between coronary plaque morphology of the left anterior descending artery and 12 months clinical outcome: the CLIMA study. Eur Heart J. 2020 Jan 14;41(3):383-391. doi: 10.1093/eurheartj/ehz520. PMID 31504405
- [Background] Di Vito L, Cattabiani MA, Paoletti G, Yoon JH, Chisari A, Gramegna M, Versaci F, Castriota F, Prati F. Comparison between intermediate and severe coronary stenoses and clinical outcomes of an OCT-guided PCI strategy. J Cardiovasc Med (Hagerstown). 2016 May;17(5):361-7. doi: 10.2459/JCM.0000000000000280. PMID 26258719
- [Background] Prati F, Romagnoli E, Burzotta F, Limbruno U, Gatto L, La Manna A, Versaci F, Marco V, Di Vito L, Imola F, Paoletti G, Trani C, Tamburino C, Tavazzi L, Mintz GS. Clinical Impact of OCT Findings During PCI: The CLI-OPCI II Study. JACC Cardiovasc Imaging. 2015 Nov;8(11):1297-305. doi: 10.1016/j.jcmg.2015.08.013. PMID 26563859
- [Background] Prati F, Di Vito L, Biondi-Zoccai G, Occhipinti M, La Manna A, Tamburino C, Burzotta F, Trani C, Porto I, Ramazzotti V, Imola F, Manzoli A, Materia L, Cremonesi A, Albertucci M. Angiography alone versus angiography plus optical coherence tomography to guide decision-making during percutaneous coronary intervention: the Centro per la Lotta contro l'Infarto-Optimisation of Percutaneous Coronary Intervention (CLI-OPCI) study. EuroIntervention. 2012 Nov 22;8(7):823-9. doi: 10.4244/EIJV8I7A125. PMID 23034247
- [Background] Witzenbichler B, Maehara A, Weisz G, Neumann FJ, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Stuckey TD, Mazzaferri EL Jr, Xu K, Parise H, Mehran R, Mintz GS, Stone GW. Relationship between intravascular ultrasound guidance and clinical outcomes after drug-eluting stents: the assessment of dual antiplatelet therapy with drug-eluting stents (ADAPT-DES) study. Circulation. 2014 Jan 28;129(4):463-70. doi: 10.1161/CIRCULATIONAHA.113.003942. Epub 2013 Nov 26. PMID 24281330
- [Background] Ahn JM, Kang SJ, Yoon SH, Park HW, Kang SM, Lee JY, Lee SW, Kim YH, Lee CW, Park SW, Mintz GS, Park SJ. Meta-analysis of outcomes after intravascular ultrasound-guided versus angiography-guided drug-eluting stent implantation in 26,503 patients enrolled in three randomized trials and 14 observational studies. Am J Cardiol. 2014 Apr 15;113(8):1338-47. doi: 10.1016/j.amjcard.2013.12.043. Epub 2014 Jan 31. PMID 24685326

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT07182799/Prot_SAP_000.pdf